CLINICAL TRIAL: NCT02290223
Title: Patient Activation to Address Chronic Pain and Opioid Management in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN-14-1928-H
Record Dates: First submitted 2014-10-27; First posted 2014-11-14 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Analgesics, Opioid; Cognitive Therapy; Behavior Therapy; Mindfulness; Psychophysiology; Biofeedback, Psychology
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Activation Group Intervention (Experimental): The experimental procedure is a behavioral based treatment model, plus usual care which is is determined by patients' individual providers, according to practice guidelines related to specific conditions.
  Interventions: Behavioral: Behavioral Based Treatment Model
- Usual Care (No Intervention): Usual care is determined by patients' individual providers, according to practice guidelines related to specific conditions.

INTERVENTIONS:
Behavioral: Behavioral Based Treatment Model — Behavioral based treatment consists of four 90 minute group sessions, one meeting per week. The sessions addressed: empowering patients to take an active role in pain management and overall health; pain management lifestyle practices; use of health information technology resources for active self-care; education on neurobiology of pain and opioids; and improving communication with providers.
  Arms: Patient Activation Group Intervention

SUMMARY:
Will a primary care-based behavioral intervention for patient activation and engagement and self-management, for patients with chronic pain who are taking opioid pain medication, result in better patient outcomes than Usual Care?

DETAILED DESCRIPTION:
Patients with chronic pain (PWCP) typically have multiple chronic conditions, and many points of contact with the health system. They can feel disempowered, and experience fragmented care and poor outcomes. PWCP report concerns about under-treatment of pain, difficulties in obtaining medication, and stigma. Prescription opioids are a very common, and controversial, pain treatment. PWCP often lack the skills and knowledge to talk to their physicians about their pain and opioid use, and to navigate the health care system. The study's aims compare the effectiveness of an innovative behavioral Patient Activation plus Usual Care (PA+UC) intervention to Usual Care (UC) only on patient-centered outcomes among PWCP. While most studies have focused on chronic opioid users, this takes an upstream approach, focusing on patients as they start regular opioid use. The overarching research question is: Can patients' increased activation improve their quality of life? With our stakeholder group of patient, clinical, and operational advisors, we propose a pragmatic, randomized trial to examine the comparative effectiveness of a group-based PA intervention in two large primary care clinics in Kaiser Permanente Northern California (KPNC). We will randomize 324 PWCP to either the PA+UC arm or UC only arm. The curriculum will cover patient activation and empowerment, how to talk to doctors about prescription opioid use, and self-management of chronic pain, including how to navigate the health care system and a patient portal. We will further develop the study questions, intervention curriculum, outcome measures, and dissemination plan with our stakeholder groups. We will examine effects over 12 months using follow-up patient interviews combined with electronic health records and a mixed effects modeling approach. Patient outcomes include patient-reported activation, quality of life, prescription opioid use, pain severity and function, patient-provider communication, patient satisfaction, knowledge of opioid use risks and benefits, self-care, including use of health information technology, and service utilization.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged 18+ who receive primary care at the Kaiser Permanente Santa Clara or San Jose Medical Center study clinic
2. Patients who have been using prescription opioids for pain at least three days per week over the past three months.47,48,60

Exclusion criteria:

1. Patients who have any other more serious comorbidity than their pain (e.g., terminal illness, active cancer, high risk for/currently with uncontrolled addictions or severe mental health issues such as psychosis), or impairing ability to engage with interventions
2. Patients who are already treated in pain clinic
3. Patients who are already treated in chemical dependency treatment
4. Patients who do not read and understand English
5. Patients planning to taper or stop taking prescription opioids in next 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia I Campbell, PhD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente, San Jose Medical Center, San Jose, California
  - Kaiser Permanente, Santa Clara Medical Center, Santa Clara, California

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] Gureje O, Simon GE, Von Korff M. A cross-national study of the course of persistent pain in primary care. Pain. 2001 May;92(1-2):195-200. doi: 10.1016/s0304-3959(00)00483-8. PMID 11323140
- [Background] Boudreau D, Von Korff M, Rutter CM, Saunders K, Ray GT, Sullivan MD, Campbell CI, Merrill JO, Silverberg MJ, Banta-Green C, Weisner C. Trends in long-term opioid therapy for chronic non-cancer pain. Pharmacoepidemiol Drug Saf. 2009 Dec;18(12):1166-75. doi: 10.1002/pds.1833. PMID 19718704
- [Background] Caudill-Slosberg MA, Schwartz LM, Woloshin S. Office visits and analgesic prescriptions for musculoskeletal pain in US: 1980 vs. 2000. Pain. 2004 Jun;109(3):514-519. doi: 10.1016/j.pain.2004.03.006. PMID 15157714
- [Background] Ballantyne JC. Pain medicine: repairing a fractured dream. Anesthesiology. 2011 Feb;114(2):243-6. doi: 10.1097/ALN.0b013e3182039f87. No abstract available. PMID 21239973
- [Background] Deyo RA, Mirza SK, Turner JA, Martin BI. Overtreating chronic back pain: time to back off? J Am Board Fam Med. 2009 Jan-Feb;22(1):62-8. doi: 10.3122/jabfm.2009.01.080102. PMID 19124635
- [Background] Dhalla IA, Persaud N, Juurlink DN. Facing up to the prescription opioid crisis. BMJ. 2011 Aug 23;343:d5142. doi: 10.1136/bmj.d5142. No abstract available. PMID 21862533
- [Background] Grady D, Berkowitz SA, Katz MH. Opioids for chronic pain. Arch Intern Med. 2011 Sep 12;171(16):1426-7. doi: 10.1001/archinternmed.2011.213. Epub 2011 Jun 13. No abstract available. PMID 21670333
- [Background] Katz MH. Long-term opioid treatment of nonmalignant pain: a believer loses his faith. Arch Intern Med. 2010 Sep 13;170(16):1422-4. doi: 10.1001/archinternmed.2010.335. No abstract available. PMID 20837826
- [Background] McLellan AT, Turner BJ. Chronic noncancer pain management and opioid overdose: time to change prescribing practices. Ann Intern Med. 2010 Jan 19;152(2):123-4. doi: 10.7326/0003-4819-152-2-201001190-00012. No abstract available. PMID 20083830
- [Background] Okie S. A flood of opioids, a rising tide of deaths. N Engl J Med. 2010 Nov 18;363(21):1981-5. doi: 10.1056/NEJMp1011512. No abstract available. PMID 21083382
- [Background] Sullivan MD. Limiting the potential harms of high-dose opioid therapy: comment on "Opioid dose and drug-related mortality in patients with nonmalignant pain". Arch Intern Med. 2011 Apr 11;171(7):691-3. doi: 10.1001/archinternmed.2011.101. No abstract available. PMID 21482847
- [Background] Von Korff M, Kolodny A, Deyo RA, Chou R. Long-term opioid therapy reconsidered. Ann Intern Med. 2011 Sep 6;155(5):325-8. doi: 10.7326/0003-4819-155-5-201109060-00011. PMID 21893626
- [Background] Chou R, Fanciullo GJ, Fine PG, Miaskowski C, Passik SD, Portenoy RK. Opioids for chronic noncancer pain: prediction and identification of aberrant drug-related behaviors: a review of the evidence for an American Pain Society and American Academy of Pain Medicine clinical practice guideline. J Pain. 2009 Feb;10(2):131-46. doi: 10.1016/j.jpain.2008.10.009. PMID 19187890
- [Background] Chou R, Fanciullo GJ, Fine PG, Adler JA, Ballantyne JC, Davies P, Donovan MI, Fishbain DA, Foley KM, Fudin J, Gilson AM, Kelter A, Mauskop A, O'Connor PG, Passik SD, Pasternak GW, Portenoy RK, Rich BA, Roberts RG, Todd KH, Miaskowski C; American Pain Society-American Academy of Pain Medicine Opioids Guidelines Panel. Clinical guidelines for the use of chronic opioid therapy in chronic noncancer pain. J Pain. 2009 Feb;10(2):113-30. doi: 10.1016/j.jpain.2008.10.008. PMID 19187889
- [Background] Papaleontiou M, Henderson CR Jr, Turner BJ, Moore AA, Olkhovskaya Y, Amanfo L, Reid MC. Outcomes associated with opioid use in the treatment of chronic noncancer pain in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2010 Jul;58(7):1353-69. doi: 10.1111/j.1532-5415.2010.02920.x. Epub 2010 Jun 1. PMID 20533971
- [Background] Sullivan MD, Von Korff M, Banta-Green C, Merrill JO, Saunders K. Problems and concerns of patients receiving chronic opioid therapy for chronic non-cancer pain. Pain. 2010 May;149(2):345-353. doi: 10.1016/j.pain.2010.02.037. Epub 2010 Mar 23. PMID 20334974
- [Background] Sullivan MD, Ballantyne JC. What are we treating with long-term opioid therapy? Arch Intern Med. 2012 Mar 12;172(5):433-4. doi: 10.1001/archinternmed.2011.2156. No abstract available. PMID 22412109
- [Background] Volkow ND, McLellan TA. Curtailing diversion and abuse of opioid analgesics without jeopardizing pain treatment. JAMA. 2011 Apr 6;305(13):1346-7. doi: 10.1001/jama.2011.369. No abstract available. PMID 21467287
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Warner M, Chen LH, Makuc DM. Increase in fatal poisonings involving opioid analgesics in the United States, 1999-2006. NCHS Data Brief. 2009 Sep;(22):1-8. PMID 19796521
- [Background] Coben JH, Davis SM, Furbee PM, Sikora RD, Tillotson RD, Bossarte RM. Hospitalizations for poisoning by prescription opioids, sedatives, and tranquilizers. Am J Prev Med. 2010 May;38(5):517-24. doi: 10.1016/j.amepre.2010.01.022. PMID 20409500
- [Background] Substance Abuse and Mental Health Services Administration, Office of Applied Studies. The DAWN Report: Trends in Emergency Department visits involving nonmedical use of narcotic pain relievers. Rockville, MD. June 18, 2010. http://www.samhsa.gov/data/2k10/DAWN016/OpioidED.htm. Accessed January 19, 2012.
- [Background] Substance Abuse and Mental Health Services Administration. Table 1.1a. Admissions aged 12 and older, by primary substance of abuse: 1999-2009. Treatment Episode Dataset (TEDS) 1999-2009. National Admissions to Substance Abuse Treatment Services. 2010. http://www.samhsa.gov/data/DASIS/teds09/TEDS2k9NTbl1.1a.htm. Accessed January 19, 2014.
- [Background] U. S. Food and Drug Administration. Questions and answers: FDA approves a Risk Evaluation and Mitigation Strategy (REMS) for Extended-Release and Long-Acting (ER/LA) opioid analgesics. Drugs. 2012. http://www.fda.gov/Drugs/DrugSafety/InformationbyDrugClass/ucm309742.htm. Updated March 1, 2013. Accessed January 17, 2014.
- [Background] U. S. Food and Drug Administration. Background on opioid REMS. Drugs. 2012. http://www.fda.gov/Drugs/DrugSafety/InformationbyDrugClass/ucm187975.htm. Updated April 22, 2013. Accessed January 17, 2014.
- [Background] Trescott CE, Beck RM, Seelig MD, Von Korff MR. Group Health's initiative to avert opioid misuse and overdose among patients with chronic noncancer pain. Health Aff (Millwood). 2011 Aug;30(8):1420-4. doi: 10.1377/hlthaff.2011.0759. PMID 21821559
- [Background] Von Korff MR. Opioids for chronic noncancer pain: as the pendulum swings, who should set prescribing standards for primary care? Ann Fam Med. 2012 Jul-Aug;10(4):302-3. doi: 10.1370/afm.1422. No abstract available. PMID 22778117
- [Background] Ballantyne JC. Patient-centered health care: are opioids a special case? Spine J. 2009 Sep;9(9):770-2. doi: 10.1016/j.spinee.2009.06.006. Epub 2009 Jul 29. No abstract available. PMID 19643676
- [Background] Frantsve LM, Kerns RD. Patient-provider interactions in the management of chronic pain: current findings within the context of shared medical decision making. Pain Med. 2007 Jan-Feb;8(1):25-35. doi: 10.1111/j.1526-4637.2007.00250.x. PMID 17244101
- [Background] Matthias MS, Parpart AL, Nyland KA, Huffman MA, Stubbs DL, Sargent C, Bair MJ. The patient-provider relationship in chronic pain care: providers' perspectives. Pain Med. 2010 Nov;11(11):1688-97. doi: 10.1111/j.1526-4637.2010.00980.x. PMID 21044259
- [Background] Matthias MS, Krebs EE, Collins LA, Bergman AA, Coffing J, Bair MJ. "I'm not abusing or anything": patient-physician communication about opioid treatment in chronic pain. Patient Educ Couns. 2013 Nov;93(2):197-202. doi: 10.1016/j.pec.2013.06.021. Epub 2013 Aug 2. PMID 23916677
- [Background] Frosch DL, May SG, Rendle KA, Tietbohl C, Elwyn G. Authoritarian physicians and patients' fear of being labeled 'difficult' among key obstacles to shared decision making. Health Aff (Millwood). 2012 May;31(5):1030-8. doi: 10.1377/hlthaff.2011.0576. PMID 22566443
- [Background] Upshur CC, Bacigalupe G, Luckmann R. "They don't want anything to do with you": patient views of primary care management of chronic pain. Pain Med. 2010 Dec;11(12):1791-8. doi: 10.1111/j.1526-4637.2010.00960.x. Epub 2010 Oct 1. PMID 21029353
- [Background] Putre L. Caring for health care's costliest patients: Aligning Forces for Equality & Robert Wood Johnson Foundation. 2014. http://www.rwjf.org/content/dam/farm/reports/issue_briefs/2014/rwjf409911. Accessed January 17, 2014
- [Background] Brumder T, Wood SB. Strategies to improve linkages between primary care and substance abuse treatment. Treatment Research Center Conference on Clinical Innovations in Substance Abuse Treatment May 19, 2012; University of California San Francisco, CA
- [Background] Weisner C, Parthasarathy S, Chi F, et al. Integrating alcohol and drug treatment with primary care: a medical home model. Treatment Research Center Conference on Clinical Innovations in Substance Abuse Treatment May 19, 2012; University of California San Francisco, CA
- [Background] Office of the National Coordinator for Health Information Technology. Policymaking, regulation, & strategy. Meaningful use. HealthIT.gov. 2013. http://www.healthit.gov/policy-researchers-implementers/meaningful-use. Accessed January 19, 2014
- [Background] Chewning B, Bylund CL, Shah B, Arora NK, Gueguen JA, Makoul G. Patient preferences for shared decisions: a systematic review. Patient Educ Couns. 2012 Jan;86(1):9-18. doi: 10.1016/j.pec.2011.02.004. Epub 2011 Apr 6. PMID 21474265
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Towle A, Godolphin W. Framework for teaching and learning informed shared decision making. BMJ. 1999 Sep 18;319(7212):766-71. doi: 10.1136/bmj.319.7212.766. No abstract available. PMID 10488010
- [Background] Driessen E, Hollon S. Motivational interviewing from a cognitive behavioral perspective. Cogn Behav Pract. 2011;18:70-73
- [Background] Rollnick S, Butler CC, Kinnersley P, Gregory J, Mash B. Motivational interviewing. BMJ. 2010 Apr 27;340:c1900. doi: 10.1136/bmj.c1900. No abstract available. PMID 20423957
- [Background] Miller WR, Rollnick S, eds. Motivational Interviewing : Preparing People for Change. 2nd ed. New York: Guildord Press; 2002
- [Background] Debar LL, Kindler L, Keefe FJ, Green CA, Smith DH, Deyo RA, Ames K, Feldstein A. A primary care-based interdisciplinary team approach to the treatment of chronic pain utilizing a pragmatic clinical trials framework. Transl Behav Med. 2012 Dec 1;2(4):523-530. doi: 10.1007/s13142-012-0163-2. Epub 2012 Aug 30. PMID 23440672
- [Background] Edlund MJ, Martin BC, Russo JE, DeVries A, Braden JB, Sullivan MD. The role of opioid prescription in incident opioid abuse and dependence among individuals with chronic noncancer pain: the role of opioid prescription. Clin J Pain. 2014 Jul;30(7):557-64. doi: 10.1097/AJP.0000000000000021. PMID 24281273
- [Background] Edlund MJ, Sullivan M, Steffick D, Harris KM, Wells KB. Do users of regularly prescribed opioids have higher rates of substance use problems than nonusers? Pain Med. 2007 Nov-Dec;8(8):647-56. doi: 10.1111/j.1526-4637.2006.00200.x. PMID 18028043
- [Background] Brown JL, Edwards PS, Atchison JW, Lafayette-Lucey A, Wittmer VT, Robinson ME. Defining patient-centered, multidimensional success criteria for treatment of chronic spine pain. Pain Med. 2008 Oct;9(7):851-62. doi: 10.1111/j.1526-4637.2007.00357.x. PMID 18950440
- [Background] Casarett D, Karlawish J, Sankar P, Hirschman K, Asch DA. Designing pain research from the patient's perspective: what trial end points are important to patients with chronic pain? Pain Med. 2001 Dec;2(4):309-16. doi: 10.1046/j.1526-4637.2001.01041.x. PMID 15102235
- [Background] Turk DC, Dworkin RH, Allen RR, Bellamy N, Brandenburg N, Carr DB, Cleeland C, Dionne R, Farrar JT, Galer BS, Hewitt DJ, Jadad AR, Katz NP, Kramer LD, Manning DC, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robinson JP, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Witter J. Core outcome domains for chronic pain clinical trials: IMMPACT recommendations. Pain. 2003 Dec;106(3):337-345. doi: 10.1016/j.pain.2003.08.001. PMID 14659516
- [Background] Greene J, Hibbard JH, Sacks R, Overton V. When seeing the same physician, highly activated patients have better care experiences than less activated patients. Health Aff (Millwood). 2013 Jul;32(7):1299-305. doi: 10.1377/hlthaff.2012.1409. PMID 23836747
- [Background] Institute of Medicine (US) Committee on Health Literacy; Nielsen-Bohlman L, Panzer AM, Kindig DA, editors. Health Literacy: A Prescription to End Confusion. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216032/ PMID 25009856
- [Background] Pain Survey Executive Summary. Massachusetts Pain Initiative. 2010. http://www.masspaininitiative.org/files/MassPI%20Pain%20Survey%20-%20Executive%20Summary%20v3.pdf. Updated August 15, 2013. Accessed January 18, 2014.
- [Background] Kline-Simon AH, Falk DE, Litten RZ, Mertens JR, Fertig J, Ryan M, Weisner CM. Posttreatment low-risk drinking as a predictor of future drinking and problem outcomes among individuals with alcohol use disorders. Alcohol Clin Exp Res. 2013 Jan;37 Suppl 1(0 1):E373-80. doi: 10.1111/j.1530-0277.2012.01908.x. Epub 2012 Jul 24. PMID 22827502
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Lu Y. Integrating primary medical care with addiction treatment: a randomized controlled trial. JAMA. 2001 Oct 10;286(14):1715-23. doi: 10.1001/jama.286.14.1715. PMID 11594896
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed. Hillsdale, NJ: Lawrence Erlbaum Associates; 1988
- [Background] Demidenko E. Sample size and optimal design for logistic regression with binary interaction. Stat Med. 2008 Jan 15;27(1):36-46. doi: 10.1002/sim.2980. PMID 17634969
- [Background] Hsieh FY, Bloch DA, Larsen MD. A simple method of sample size calculation for linear and logistic regression. Stat Med. 1998 Jul 30;17(14):1623-34. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-s. PMID 9699234
- [Background] Sullivan MD, Edlund MJ, Zhang L, Unutzer J, Wells KB. Association between mental health disorders, problem drug use, and regular prescription opioid use. Arch Intern Med. 2006 Oct 23;166(19):2087-93. doi: 10.1001/archinte.166.19.2087. PMID 17060538
- [Background] Weisner C, Mertens J, Parthasarathy S, Moore C, Hunkeler EM, Hu T, Selby JV. The outcome and cost of alcohol and drug treatment in an HMO: day hospital versus traditional outpatient regimens. Health Serv Res. 2000 Oct;35(4):791-812. PMID 11055449
- [Background] Green CA, Perrin NA, Polen MR, Leo MC, Hibbard JH, Tusler M. Development of the Patient Activation Measure for mental health. Adm Policy Ment Health. 2010 Jul;37(4):327-33. doi: 10.1007/s10488-009-0239-6. Epub 2009 Aug 29. PMID 19728074
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Mosen DM, Schmittdiel J, Hibbard J, Sobel D, Remmers C, Bellows J. Is patient activation associated with outcomes of care for adults with chronic conditions? J Ambul Care Manage. 2007 Jan-Mar;30(1):21-9. doi: 10.1097/00004479-200701000-00005. PMID 17170635
- [Background] Schmittdiel J, Mosen DM, Glasgow RE, Hibbard J, Remmers C, Bellows J. Patient Assessment of Chronic Illness Care (PACIC) and improved patient-centered outcomes for chronic conditions. J Gen Intern Med. 2008 Jan;23(1):77-80. doi: 10.1007/s11606-007-0452-5. Epub 2007 Nov 21. PMID 18030539
- [Background] Camacho FT, Feldman SR, Balkrishnan R, Kong MC, Anderson RT. Validation and reliability of 2 specialty care satisfaction scales. Am J Med Qual. 2009 Jan-Feb;24(1):12-8. doi: 10.1177/1062860608326416. Epub 2008 Dec 5. PMID 19060254
- [Background] PROMIS Network Center. PROMIS (Patient Reported Outcome Measurement Information System). USA.gov. http://www.nihpromis.org/?AspxAutoDetectCookieSupport=1#3. Accessed January 18, 2014
- [Background] Broderick JE, DeWitt EM, Rothrock N, Crane PK, Forrest CB. Advances in Patient-Reported Outcomes: The NIH PROMIS((R)) Measures. EGEMS (Wash DC). 2013 Aug 2;1(1):1015. doi: 10.13063/2327-9214.1015. eCollection 2013. PMID 25848562
- [Background] Hinchcliff M, Beaumont JL, Thavarajah K, Varga J, Chung A, Podlusky S, Carns M, Chang RW, Cella D. Validity of two new patient-reported outcome measures in systemic sclerosis: Patient-Reported Outcomes Measurement Information System 29-item Health Profile and Functional Assessment of Chronic Illness Therapy-Dyspnea short form. Arthritis Care Res (Hoboken). 2011 Nov;63(11):1620-8. doi: 10.1002/acr.20591. PMID 22034123
- [Background] Beaumont JL, Cella D, Phan AT, Choi S, Liu Z, Yao JC. Comparison of health-related quality of life in patients with neuroendocrine tumors with quality of life in the general US population. Pancreas. 2012 Apr;41(3):461-6. doi: 10.1097/MPA.0b013e3182328045. PMID 22422138
- [Background] Flynn KE, Reeve BB, Lin L, Cyranowski JM, Bruner DW, Weinfurt KP. Construct validity of the PROMIS(R) sexual function and satisfaction measures in patients with cancer. Health Qual Life Outcomes. 2013 Mar 11;11:40. doi: 10.1186/1477-7525-11-40. PMID 23497200
- [Background] Flynn KE, Lin L, Cyranowski JM, Reeve BB, Reese JB, Jeffery DD, Smith AW, Porter LS, Dombeck CB, Bruner DW, Keefe FJ, Weinfurt KP. Development of the NIH PROMIS (R) Sexual Function and Satisfaction measures in patients with cancer. J Sex Med. 2013 Feb;10 Suppl 1(0 1):43-52. doi: 10.1111/j.1743-6109.2012.02995.x. PMID 23387911
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Obradovic M, Lal A, Liedgens H. Validity and responsiveness of EuroQol-5 dimension (EQ-5D) versus Short Form-6 dimension (SF-6D) questionnaire in chronic pain. Health Qual Life Outcomes. 2013 Jul 1;11:110. doi: 10.1186/1477-7525-11-110. PMID 23815777
- [Background] Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007 Aug;67(3):333-42. doi: 10.1016/j.pec.2007.05.005. Epub 2007 Jun 18. PMID 17574367
- [Background] Mertens JR, Flisher AJ, Satre DD, Weisner CM. The role of medical conditions and primary care services in 5-year substance use outcomes among chemical dependency treatment patients. Drug Alcohol Depend. 2008 Nov 1;98(1-2):45-53. doi: 10.1016/j.drugalcdep.2008.04.007. Epub 2008 Jun 20. PMID 18571875
- [Background] Von Korff M, Saunders K, Thomas Ray G, Boudreau D, Campbell C, Merrill J, Sullivan MD, Rutter CM, Silverberg MJ, Banta-Green C, Weisner C. De facto long-term opioid therapy for noncancer pain. Clin J Pain. 2008 Jul-Aug;24(6):521-7. doi: 10.1097/AJP.0b013e318169d03b. PMID 18574361
- [Result] Bernabeo E, Holmboe ES. Patients, providers, and systems need to acquire a specific set of competencies to achieve truly patient-centered care. Health Aff (Millwood). 2013 Feb;32(2):250-8. doi: 10.1377/hlthaff.2012.1120. PMID 23381517
- [Derived] Does MB, Adams SR, Kline-Simon AH, Marino C, Charvat-Aguilar N, Weisner CM, Rubinstein AL, Ghadiali M, Cowan P, Young-Wolff KC, Campbell CI. A patient activation intervention in primary care for patients with chronic pain on long term opioid therapy: results from a randomized control trial. BMC Health Serv Res. 2024 Jan 22;24(1):112. doi: 10.1186/s12913-024-10558-3. PMID 38254073

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Activation Group Intervention: The experimental procedure is a behavioral based treatment model, structured in the form of four group sessions, one meeting per week plus usual care which is is determined by patients' individual providers, according to practice guidelines related to specific conditions.
  Behavioral Based Treatment Model: The experimental procedure is a behavioral based treatment model, structured in the form of four group sessions, one meeting per week.
Period: Baseline
Arm/Group | Patient Activation Group Intervention | Usual Care
Started | 189 | 187
Completed | 189 | 187
Not Completed | 0 | 0
Period: 6 Months
Arm/Group | Patient Activation Group Intervention | Usual Care
Started | 189 | 187
Completed | 173 | 181
Not Completed | 16 | 6
Not completed — Lost to Follow-up | 9 | 6
Not completed — Withdrawal by Subject | 5 | 0
Not completed — deceased (not related to study) | 2 | 0
Period: 12 Months
Arm/Group | Patient Activation Group Intervention | Usual Care
Started | 182 (All participants were contacted at 12 mo, unless deceased or withdrawn (n=7).) | 187 (All participants were contacted at 12 mo, unless deceased or withdrawn (n=0).)
Completed | 166 | 176
Not Completed | 16 | 11
Not completed — Lost to Follow-up | 16 | 10
Not completed — Refusal | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were 376 enrolled in study and 189 assigned to intervention arm and 187 to usual care at baseline appointment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Activation Group Intervention | Usual Care | Total
Number analyzed (Participants) | 189 | 187 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (13.7) | 60.7 (12.4) | 59.8 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 105 | 219
  Male | 75 | 82 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 37 | 73
  Not Hispanic or Latino | 153 | 150 | 303
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 141 | 139 | 280
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 23 | 22 | 45
Patient Activation Measure [Mean (Standard Deviation); unit: units on a scale] — Patient Activation Measure (PAM) is a 13-item validated instrument for measuring patient beliefs, knowledge, and confidence for engaging in a wide range of health behaviors.The PAM-13 is measured on a 1-100 scale, with higher score representing higher level of activation.
  units on a scale | 65.8 (15.0) | 65.2 (15.9) | 65.5 (15.4)
Pain intensity [Mean (Standard Deviation); unit: units on a scale] — PROMIS pain intensity question ("How would you rate your pain, on average?") is used to measure pain level. Average raw scores are reported on scale 1-10, with 1=no pain to 10= worst imaginable.
  units on a scale | 6.7 (1.4) | 6.7 (1.6) | 6.7 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation
Description: The Patient Activation Measure (PAM) is a 13-item instrument for measuring patient beliefs, knowledge and confidence for engaging in a wide range of health behaviors.Each item is rated 1-4 (strongly disagree =1 to strongly agree=4) and a total raw score is generated (0-52). Raw scores are converted to activation scores using a published conversion table. PAM scores are reported on a 1-100 scale, with higher scores associated with positive health outcomes such as participation in health care and treatment adherence.
Time Frame: Baseline and 6 and 12 months post randomization
Population: Due to the small number of participants who withdrew, or were lost to follow up, the number of participants interviewed at 6 months and 12 months is lower than number at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 65.8 (15.0) | 65.2 (15.9)
  6 months: number analyzed (Participants) | 173 | 181
  6 months | 67.3 (13.8) | 67.7 (14.5)
  12 months: number analyzed (Participants) | 166 | 176
  12 months | 67.7 (14.8) | 66.6 (14.0)

2. Secondary Outcome: Quality of Life: Physical Health
Description: The PROMIS Global Health score was used to assess general perceptions of health and quality of life. The 10 items that comprise the Quality of Life scale are reported as two dimensions, mental health and physical health. Raw scores for PROMIS Global Physical Health were converted to standardized T-scores using published conversion tables.T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score always represents more of the concept being measured. Thus, a person who has T-score of 60 is one standard deviation better (more healthy) than the general population.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
T score
  baseline | 38.3 (6.3) | 38.2 (6.1)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 40.2 (6.7) | 39.9 (7.0)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 40.9 (7.6) | 39.0 (6.3)

3. Secondary Outcome: Quality of Life: Mental Health
Description: The PROMIS Global Health score was used to assess general perceptions of health and quality of life. The 10 items that comprise the Quality of Life scale are reported as two dimensions, mental health and physical health. Raw scores for PROMIS Global Mental Health were converted to standardized T-scores using published conversion tables.T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score always represents more of the concept being measured. Thus, a person who has T-score of 60 is one standard deviation better (more healthy) than the general population.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
T score
  baseline | 45.8 (9.4) | 45.1 (8.3)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 47.4 (8.1) | 46.9 (8.3)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 47.8 (8.0) | 46.2 (7.8)

4. Secondary Outcome: Overall Health
Description: The Patient-Reported Outcome Measurement Information System (PROMIS) Global Health instrument is a system of highly reliable, and precise measures of patient-reported outcomes in physical and mental health and social well-being. Measure of overall health is based on a single item/rating: "In general, would you say your health is:". Answers are reported on scale 1-5, with 1=poor to 5=excellent. Average raw scores are reported, with higher scores reflecting higher functioning.
Time Frame: Baseline and 6 and 12 months post randomization
Population: Due to the small number of participants who withdrew, or lost to follow up, the number of participants interviewed at 6/12 months is lower than number at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 2.7 (0.9) | 2.6 (0.9)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 2.8 (0.9) | 2.5 (0.9)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 2.7 (0.9) | 2.4 (0.9)

5. Secondary Outcome: PHQ-9 Depression
Description: Depression was measured using the Patient Health Questionnaire-9 (PHQ-9), a reliable and well validated instrument. Mean scores are reported in range 0-27, with higher score indicating severity of depression: mild (5-9), moderate (10-14), moderately severe (15-19) and over 20 indicating severe depression.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
score
  baseline | 6.7 (5.3) | 7.0 (5.3)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 5.6 (5.1) | 6.2 (5.6)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 5.5 (4.8) | 6.2 (4.7)

6. Secondary Outcome: Satisfaction With Care
Description: Satisfaction with primary care provider is reported on a scale from 1-10, where "1" is the worst possible care and "10" is the best possible care. Mean scores are reported, and higher scores indicates more satisfaction with care.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 8.6 (1.8) | 8.6 (1.7)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 8.5 (1.8) | 8.6 (1.8)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 8.7 (1.7) | 8.5 (1.8)

7. Secondary Outcome: Opioid Misuse SOAPP
Description: The Screener and Opioid Assessment for Patients in Pain (SOAPP-5) is a 5 item survey used to identify aberrant behaviors related to long-term opioid treatment. Each item is rated 0 to 4 (with 0=never and 4=very often); ratings are added for all 5 items resulting in a range of possible scores 0-20. A higher score indicates greater risk for patients on long term opioids, and a score of => 4 is considered positive. Results reported are the number and % of participants who score => 4.
Time Frame: Baseline and 6 and 12 months post randomization
Population: The numbers at 6/12 months are lower than at baseline due to lost to follow up/withdrawals. In addition, the denominators for 6/12 month SOAPP are lower than other outcomes because questions were ONLY asked if participants took opioids at 6/12 (therefore, 36 excluded at 6 months, n=19 INT, n=17 UC, and 44 excluded at 12 months, n=25 INT, n=19 UC).
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  baseline | 48 | 59
  6 months: number analyzed (Participants) | 154 | 164
  6 months | 28 | 28
  12 months: number analyzed (Participants) | 141 | 157
  12 months | 25 | 23

8. Secondary Outcome: Opioid Misuse COMM
Description: The Current Opioid Misuse Measure (COMM) is used to identify aberrant behaviors related to long-term opioid treatment. It is a clinical screening tool for monitoring patients for opioid overuse and misuse in six areas. The COMM contains 17 items with total score range of 0-68, and a score of 9 or greater is considered positive. It uses a low cut off value as it is intended to over-identify misuse. Results reported are the number and % of participants who score => 9.
Time Frame: Baseline and 6 and 12 months post randomization
Population: The numbers at 6/12 months are lower than at baseline due to lost to follow up/withdrawals. In addition, the denominators for 6/12 month COMM are lower than other outcomes because questions were ONLY asked if participants took opioids at 6/12 (therefore, 36 excluded at 6 months, n=19 INT, n=17 UC, and 44 excluded at 12 months, n=25 INT, n=19 UC).
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  baseline | 57 | 68
  6 months: number analyzed (Participants) | 154 | 164
  6 months | 22 | 25
  12 months: number analyzed (Participants) | 141 | 157
  12 months | 14 | 22

9. Secondary Outcome: Pain Coping
Description: The 42-item Chronic Pain Coping Inventory (CPCI) is used to assess behavioral and cognitive pain coping strategies. It contains 8 subscales: Guarding, Resting, Asking for Assistance, Relaxation, Task Persistence, Exercising/Stretching, Coping Self-Statements, and Seeking Social Support. For each subscale, patients were asked the number of days (0-7 days) he/she performed each task (4-7 tasks). The mean score for each subscale is reported, with possible range of scores 0-7. The CPCI was developed to assess the behavioral coping strategies that are taught and encouraged during treatment (eg, relaxation, exercising, task persistence), ones that are discouraged (eg, guarding, resting, asking for assistance), and one neutral strategy (seeking social support). Active strategies are defined as adaptive coping responses (eg, staying busy or active), and higher scores are associated with positive coping.
Time Frame: 6 and 12 months post randomization
Population: For brevity purposes, the baseline values are not included in the table (n=189 intervention and n=187usual care). There were 354 participants included in the 6 mo analysis (n=173 intervention and n=181 usual care) and 342 participants in 12 mo analysis (n=166 intervention and n=176 usual care).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 173 | 181
units on a scale
  6 month Guarding | 3.6 (1.9) | 3.7 (1.8)
  12 month Guarding: number analyzed (Participants) | 166 | 176
  12 month Guarding | 3.4 (2.0) | 3.6 (2.0)
  6 month Resting | 4.3 (1.8) | 3.9 (2.0)
  12 month Resting: number analyzed (Participants) | 166 | 176
  12 month Resting | 3.8 (1.7) | 3.8 (2.0)
  6 month Asking for assistance | 2.5 (2.2) | 2.7 (2.3)
  12 month Asking for assistance: number analyzed (Participants) | 166 | 176
  12 month Asking for assistance | 2.5 (2.3) | 2.5 (2.4)
  6 month Relaxation | 3.0 (1.8) | 2.5 (2.0)
  12 month Relaxation: number analyzed (Participants) | 166 | 176
  12 month Relaxation | 2.9 (2.0) | 2.3 (1.9)
  6 month Task persistence | 4.8 (1.8) | 4.7 (1.7)
  12 month Task persistence: number analyzed (Participants) | 166 | 176
  12 month Task persistence | 4.9 (1.8) | 4.7 (1.8)
  6 month Exercise/stretching | 3.2 (1.9) | 3.1 (2.0)
  12 month Exercise/stretching: number analyzed (Participants) | 166 | 176
  12 month Exercise/stretching | 3.3 (2.1) | 2.8 (2.0)
  6 month Seeking social support | 2.9 (2.1) | 2.8 (2.1)
  12 month Seeking social support: number analyzed (Participants) | 166 | 176
  12 month Seeking social support | 3.0 (2.1) | 2.8 (2.2)
  6 month Coping self-statements | 4.5 (2.0) | 4.4 (2.1)
  12 month Coping self-statements: number analyzed (Participants) | 166 | 176
  12 month Coping self-statements | 4.5 (2.1) | 4.4 (2.1)

10. Secondary Outcome: Self-Efficacy
Description: Pain Self-Efficacy Questionnaire (PSEQ) is an established 10-item measure of pain self-efficacy that is widely used in clinical settings to assess confidence in one's ability to work and lead a normal life despite pain. Each item is rated on a 7-point scale with 0= not at all confident and 6=extremely confident. A total score is calculated by summing the scores for each of 10 items, yielding max score of 60. A higher score indicates higher self-efficacy.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 34.1 (13.3) | 35.7 (13.4)
  6 months: number analyzed (Participants) | 173 | 181
  6 months | 40.2 (12.6) | 39.6 (13.1)
  12 months: number analyzed (Participants) | 166 | 176
  12 months | 42.3 (11.8) | 40.0 (11.7)

11. Secondary Outcome: Pain Intensity
Description: Measured with the Patient-Reported Outcome Measurement Information System (PROMIS) Global Health instrument. PROMIS is a system of highly reliable, and precise measures of patient-reported outcomes in physical and mental health and social well-being. Pain intensity is assessed using a single item ("How would you rate your pain, on average?"). The average raw score is reported on scale 1-10, with 1=no pain to 10= worst imaginable.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 6.7 (1.4) | 6.7 (1.6)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 5.9 (1.8) | 5.9 (1.9)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 5.8 (2.1) | 6.1 (1.7)

12. Secondary Outcome: Function: Everyday Physical Activities
Description: The Patient-Reported Outcome Measurement Information System (PROMIS) Global Health instrument is a system of highly reliable, and precise measures of patient-reported outcomes in physical and mental health and social well-being. This function domain is based on a single item: "To what extent are you able to carry out your everyday physical activities such as walking, climbing stairs, carrying groceries, or moving a chair?" Answers are reported on scale 1-5, with 1=not at all to 5=completely. Average raw scores are reported, with higher scores reflecting higher functioning.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 3.4 (1.0) | 3.3 (1.0)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 3.4 (1.1) | 3.4 (1.1)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 3.6 (1.1) | 3.3 (1.1)

13. Secondary Outcome: Function: Social Activities and Roles
Description: The Patient-Reported Outcome Measurement Information System (PROMIS) Global Health instrument is a system of highly reliable, and precise measures of patient-reported outcomes in physical and mental health and social well-being. This function domain is based on a single item: "In general, please rate how well you carry out your usual social activities and roles. (This includes activities at home, at work and in your community, and responsibilities as a parent, child, spouse, employee, friend, etc.)" Answers are reported on scale 1-5, with 1=poor to 5=excellent. Average raw scores are reported, with higher scores reflecting higher functioning.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 3.3 (1.1) | 3.1 (1.1)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 3.3 (0.9) | 3.3 (1.0)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 3.3 (1.0) | 3.1 (0.9)

14. Secondary Outcome: Patient Provider Communication
Description: The Communication Assessment Tool (CAT) measures patients' perceptions of physician performance with regard to communication and interpersonal skills. It is a 14-item instrument that asks respondents to rate their primary primary care physician based on the last couple of visits. The answers are reported using a 5-point rating scale, with 1=poor to 5=excellent. Average scores are reported.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 4.3 (0.8) | 4.2 (0.9)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 4.2 (1.0) | 4.2 (1.0)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 4.3 (1.0) | 4.2 (1.0)

15. Secondary Outcome: Patient Provider Interactions
Description: The Perceived Efficacy in Patient-Physician Interactions Questionnaire (PEPPI) is used to measure patients' self-efficacy in obtaining medical information and attention to their medical concerns from physicians.Ten questions are measured on a scale from 1 (not at all confident) to 5 (very confident) and the range of possible scores is 10-50. Average scores are reported, with higher score reflecting more confidence in interacting with his/her physician.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
units on a scale
  baseline | 43.4 (7.8) | 43.3 (7.9)
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 44.9 (6.6) | 44.7 (6.9)
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 45.6 (6.8) | 45.9 (5.6)

16. Secondary Outcome: Health Care Utilization Service Visits (EHR)
Description: Primary care services (number of non-urgent outpatient visits) and acute care services (number of emergency room (ER) visits and inpatient stays) within KPNC as extracted from the electronic health records are reported. Average number of visits are reported for 6 month period prior to baseline, for 3 months prior to 6 month interview, and 6 months prior to 12 month interview. For all three time periods, active membership in Kaiser health plan is required for 4 of 6 months, and 3 of 3 months for the 3-month period used in 6 month analysis.
Time Frame: Baseline and 6 and 12 months post randomization
Population: EHR data were extracted for all study participants who remained active Kaiser members in the follow-up period, regardless of whether they completed the follow-up surveys or not. Due to incomplete membership in the follow-up period, 13 people were excluded from the 6-month EHR outcomes, and 16 people were excluded from the 12-month EHR outcomes.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
visits
  baseline primary care visits | 2.9 (3.3) | 2.7 (2.5)
  6 month primary care visits: number analyzed (Participants) | 181 | 182
  6 month primary care visits | 1.2 (1.6) | 1.2 (1.5)
  12 month primary care visits: number analyzed (Participants) | 178 | 182
  12 month primary care visits | 2.9 (3.0) | 2.7 (3.5)
  baseline ER visits | 0.4 (0.7) | 0.5 (1.9)
  6 month ER visits: number analyzed (Participants) | 181 | 182
  6 month ER visits | 0.1 (0.4) | 0.2 (0.5)
  12 month ER visits: number analyzed (Participants) | 178 | 182
  12 month ER visits | 0.3 (0.8) | 0.3 (0.9)
  baseline Inpatient stays | 0.1 (0.4) | 0.2 (0.5)
  6 month Inpatient stays: number analyzed (Participants) | 181 | 182
  6 month Inpatient stays | 0.0 (0.3) | 0.0 (0.2)
  12 month Inpatient stays: number analyzed (Participants) | 178 | 182
  12 month Inpatient stays | 0.1 (0.3) | 0.1 (0.3)

17. Secondary Outcome: Health Care Utilization Portal Use (EHR)
Description: Use of Kaiser's online portal is extracted from electronic health record. Results are reported as number and % of patients who used the portal during specified time periods: 1) 6 month period prior to baseline, 2) 3 months prior to 6 month interview, and 3) 6 months prior to 12 month interview. For all three time periods, active membership in Kaiser health plan is required for 4 of 6 months, and 3 of 3 months for the 3-month period used in 6 month analysis.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  baseline | 168 | 157
  6 month: number analyzed (Participants) | 181 | 182
  6 month | 164 | 152
  12 month: number analyzed (Participants) | 178 | 182
  12 month | 160 | 156

18. Secondary Outcome: Use of Online Health and Wellness Resources (Self-reported)
Description: Use of Kaiser's online portal (kp.org) was reported by participants on questionnaire at baseline, 6 and 12 months. Participants were asked different ways in which portal was used, and if they used kp.org's health and wellness resources (healthy lifestyle programs, wellness coaching, audio podcasts, recipe blogs, tools/calculators, videos). Results reported here are number and % of patients who reported using Kaiser's online health and wellness resources during specified time period ("ever" at baseline, and "past 6 months" at 6/12 months).
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  baseline | 47 | 42
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 68 | 50
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 76 | 50

19. Secondary Outcome: Attendance at Health Education Classes (Self-reported)
Description: Attendance at Kaiser's health education classes was reported by participants on questionnaire at baseline, 6 and 12 months. Results are reported as number and % of patients who attended health education class during specified time period ("ever" at baseline, and "past 6 months" at 6/12 months).
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  baseline | 113 | 108
  6 month: number analyzed (Participants) | 173 | 181
  6 month | 22 | 20
  12 month: number analyzed (Participants) | 166 | 176
  12 month | 22 | 18

20. Secondary Outcome: Prescription Opioid Use (EHR)
Description: Opioid prescription dispensations were extracted from electronic health records and converted into morphine milligram equivalent (MME), by multiplying the quantity of each prescription by the strength of prescription (milligrams of opioid/unit dispensed). The resulting product is then multiplied by the conversion factor for MMEs. We calculated the average daily MME dispensed for the relevant time periods. Results are reported for 3 time periods: 1) 6 months prior to baseline, 2) 3 months prior to 6 month interview, and 3) 6 months prior to 12 month interview. For all 3 time periods, active membership in Kaiser health plan is required for 4 of 6 months, and 3 of 3 months for the 3-month period used in 6 month analysis.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
MME
  Baseline | 35.8 (68.9) | 32.1 (43.8)
  6 months: number analyzed (Participants) | 181 | 182
  6 months | 30.4 (64.3) | 28.2 (35.5)
  12 months: number analyzed (Participants) | 178 | 182
  12 months | 28.0 (70.7) | 25.3 (32.9)

21. Secondary Outcome: Pain Management Strategies- Mindfulness, Meditation and Relaxation
Description: Participants were asked to identify which of the following they were currently using to manage their pain: opioid medication prescribed by a doctor; non-opioid medication prescribed by a doctor; over the counter medication; complementary/alternative medicine; meditation, relaxation, or mindfulness practice; pain classes or therapy; massage or other bodywork; exercise, stretching or physical therapy; or other. Results are reported as number and percent of participants who endorsed "mindfulness, meditation and relaxation". Only the outcomes with significant differences between two arms at 6 and/or 12 months are reported.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  Baseline | 64 | 50
  6 months: number analyzed (Participants) | 173 | 181
  6 months | 75 | 45
  12 months: number analyzed (Participants) | 166 | 176
  12 months | 61 | 34

22. Secondary Outcome: Pain Management Strategies- Exercise, Stretching or Physical Therapy
Description: Participants were asked to identify which of the following they were currently using to manage their pain: opioid medication prescribed by a doctor; non-opioid medication prescribed by a doctor; over the counter medication; complementary/alternative medicine; meditation, relaxation, or mindfulness practice; pain classes or therapy; massage or other bodywork; exercise, stretching or physical therapy; or other. Results are reported as number and percent of participants who endorsed "exercise, stretching or physical therapy". Only the outcomes with significant differences between two arms at 6 and/or 12 months are reported.
Time Frame: Baseline and 6 and 12 months post randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  Baseline | 108 | 95
  6 months: number analyzed (Participants) | 173 | 181
  6 months | 120 | 123
  12 months: number analyzed (Participants) | 166 | 176
  12 months | 127 | 100

23. Secondary Outcome: Goals for Opioid Use at Baseline
Description: Participants were asked at baseline about their long-term goals for using prescription opioids for pain management. Results are presented as number and percent who wanted to stay the same/increase use, and number and percent who wanted to decrease or stop use of prescription opioids.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  Stay same/increase use | 67 | 76
  Decrease/stop use | 122 | 111

24. Secondary Outcome: Met Baseline Goals for Opioid Use at 6 and 12 Months
Description: Participants were asked at 6 and12 months to what extent they felt they met goals for opioid use stated at baseline. Results are presented as number and percent who reported "to a great extent"/"somewhat", vs. "very little"/"not al all".
Time Frame: 6 and 12 months post-randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  6 months: number analyzed (Participants) | 173 | 181
  6 months: To a great extent/somewhat | 131 | 132
  6 months: Very little/not at all | 42 | 49
  6 months: missing | 0 | 0
  12 months: number analyzed (Participants) | 166 | 176
  12 months: To a great extent/somewhat | 131 | 127
  12 months: Very little/not at all | 35 | 45
  12 months: missing | 0 | 4

25. Secondary Outcome: Substance Use
Description: Participants were asked about 9 categories of substance use in past 3 months, based on NIDA-modified Alcohol, Smoking and Substance Involvement Screening Test (ASSIST). Results are reported as number and percent for three categories: prescription/street opioids, cannabis and sedatives/sleeping pills. Remaining categories (cocaine, methamphetamines, stimulants, inhalants) were collapsed into "other" category.
Time Frame: Baseline and 6 and 12 month post-randomization
Population: Due to the small number of participants who withdrew, or lost to follow up, the number of participants interviewed at 6/12 months is lower than number at baseline. Categories do not add up to number analyzed because answer were "check all that apply" and multiple answers per respondent were allowed.
Measure: Number; unit: participants who used given substance
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
participants who used given substance
  Baseline substance use : Cannabis | 23 | 29
  Baseline substance use : Sedatives/sleeping pills | 53 | 51
  Baseline substance use : Opioids | 160 | 173
  Baseline substance use : Other | 11 | 10
  6 month substance use : Cannabis: number analyzed (Participants) | 173 | 181
  6 month substance use : Cannabis | 19 | 20
  6 month substance use : Sedatives/sleeping pills: number analyzed (Participants) | 173 | 181
  6 month substance use : Sedatives/sleeping pills | 35 | 35
  6 month substance use : Opioids: number analyzed (Participants) | 173 | 181
  6 month substance use : Opioids | 135 | 147
  6 month substance use : Other: number analyzed (Participants) | 173 | 181
  6 month substance use : Other | 3 | 1
  12 month substance use : Cannabis: number analyzed (Participants) | 166 | 176
  12 month substance use : Cannabis | 22 | 17
  12 month substance use : Sedatives/sleeping pills: number analyzed (Participants) | 166 | 176
  12 month substance use : Sedatives/sleeping pills | 51 | 43
  12 month substance use : Opioids: number analyzed (Participants) | 166 | 176
  12 month substance use : Opioids | 132 | 147
  12 month substance use : Other: number analyzed (Participants) | 166 | 176
  12 month substance use : Other | 6 | 2

26. Secondary Outcome: Alcohol Use
Description: The number and percent of participants who report "heavy drinking" in past 3 months are reported at baseline and 6 and 12 months. Heavy drinking is defined as 5+ drinks per day or 15+ drinks per week for males under age 65, and 4+ drinks per day or 8+ drinks per week for females and males over age 65.
Time Frame: Baseline and 6 and 12 months post-randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  baseline | 11 | 10
  6 months: number analyzed (Participants) | 173 | 181
  6 months | 8 | 9
  12 months: number analyzed (Participants) | 166 | 176
  12 months | 8 | 8

27. Secondary Outcome: Tobacco Use
Description: Participants were asked how many days they had smoked cigarettes in past 30 days at baseline, 6 and 12 months. Results are reported as number and percent who reported they smoked cigarettes on at least one day in past 30 days.
Time Frame: Baseline and 6 and 12 months post-randomization
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Activation Group Intervention | Usual Care
Number analyzed (Participants) | 189 | 187
Participants
  Baseline | 26 | 27
  6 months: number analyzed (Participants) | 173 | 181
  6 months | 17 | 24
  12 months: number analyzed (Participants) | 166 | 176
  12 months | 15 | 18

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for each participant between the date of their baseline interview and the date of their 12 month follow up interview.
Description: The electronic medical records for all study participants were reviewed during the period of active participation (between baseline interview and 12 month follow up interview). All deaths and hospitalizations were identified, discharge notes were reviewed and reason for death/hospitalizations were categorized. An Independent Safety Monitor reviewed records and determined that no serious adverse events or mortalities were related in any way to the conduct of the study.
Arm/Group | Patient Activation Group Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/189 | 1/187
Serious Adverse Events (participants affected / at risk) | 16/189 | 26/187
Other Adverse Events (participants affected / at risk) | 0/189 | 0/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Activation Group Intervention (N=189) | Usual Care (N=187)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Diastolic heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure due to pulmonary hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia repair (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic pain (General disorders) | 0 (0) | 1 (1)
Opioid withdrawal (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Post surgery Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Meningocephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Normal delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastic bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthoplasty (Surgical and medical procedures) | 3 (3) | 1 (1)
Joint fusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 2 (2) | 5 (5)
Laminotomy (Surgical and medical procedures) | 2 (2) | 2 (2)
Shoulder arthoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Left leg ischemia (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT02290223/ICF_000.pdf
  • Study Protocol (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT02290223/Prot_001.pdf
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT02290223/SAP_002.pdf